CLINICAL TRIAL: NCT00529568
Title: Randomised, Placebo-controlled, Multi-centre Study to Assess the Efficacy and Safety of Eltrombopag in Thrombocytopenic Subjects With Hepatitis C Virus (HCV) Infection Who Are Otherwise Eligible to Initiate Antiviral Therapy (Peginterferon Alfa-2b Plus Ribavirin)
Brief Title: Eltrombopag To Initiate And Maintain Interferon Antiviral Treatment To Benefit Subjects With Hepatitis C Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPL108390
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-03

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C; ribavirin; Hepatitis C-related thrombocytopenia; thrombopoietin; peginterferon alfa-2b; platelets
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- eltrombopag (Experimental): active treatment arm
  Interventions: Drug: eltrombopag
- placebo (Placebo Comparator): placebo control arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eltrombopag — double-blind active treatment daily oral administation at dose of 25, 50, 75, or 100 mg
  Arms: eltrombopag
Drug: placebo — double-blind matched placebo control daily oral administration
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the ability of eltrombopag to maintain a platelet count sufficient to facilitate initiation of antiviral therapy, to minimise antiviral therapy dose reductions and to avoid permanent discontinuation of antiviral therapy. The clinical benefit of eltrombopag will be measured by the proportion of subjects who are able to achieve a Sustained Virological Response (SVR).

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects, >18 years Evidence of chronic hepatitis C virus (HCV) infection Subjects who are appropriate candidates for peginterferon (pegIFN) and ribavirin antiviral therapy A platelet count of <75,000/mcL Haemoglobin >11.0g/dL for men or >10.0g/dL for women Absolute neutrophil count (ANC) >750/mm3 and no history of infections associated with neutropenia Creatinine clearance >50mL/minute All fertile males and females must use two forms of effective contraception between them during treatment and during the 24 weeks after treatment end Subject is able to understand, consent and comply with protocol requirements and instructions and is likely to complete the study as planned

Exclusion criteria:

Non-responders to previous treatment with pegIFN and ribavirin who failed to achieve a sustained virologic response (SVR) for reasons other than thrombocytopenia, despite an optimal course (dose and duration) of combination therapy with pegIFN and ribavirin Decompensated liver disease, e.g. Child-Pugh score >6 or history of ascites or hepatic encephalopathy or current evidence of ascites Known hypersensitivity, intolerance or allergy to interferon (IFN), ribavirin, eltrombopag or any of their ingredients Serious cardiac, cerebrovascular, or pulmonary disease that would preclude treatment with pegIFN and ribavirin

Subjects with a history of any one of the following:

Suicide attempt or hospitalisation for depression in the past 5 years Any current severe or poorly controlled psychiatric disorder

The following subjects are eligible for study participation, but must be assessed and followed (if recommended) by a mental health professional:

* Subjects who have had a severe or poorly controlled psychiatric disorder more than 6 months ago but less than 5 years ago
* Seizure disorder that has not been well controlled History of clinically significant bleeding from oesophageal or gastric varices Subjects with haemoglobinopathies, e.g. sickle cell anaemia, thalassemia major Any prior history of arterial or venous thrombosis AND two or more of the following risk factors: hereditary thrombophilic disorders (e.g. Factor V Leiden, ATIII deficiency, etc), hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension or cancer Pre-existing cardiac disease (New York Heart Association (NYHA) Grade III/IV), or arrhythmias known to involve the risk of thromboembolic events, or corrected QT interval (QTc) >450 msec Evidence of hepatocellular carcinoma Laboratory evidence of infection with human immunodeficiency virus (HIV) or active Hepatitis B Virus (HBV) infection Any disease condition associated with active bleeding or requiring anticoagulation with heparin or warfarin Therapy with any anti-neoplastic or immuno-modulatory treatment <6 months prior to the first dose of eltrombopag.

Subjects who have had a malignancy diagnosed and/or treated within the past 5 years, except for subjects with localised basal or squamous cell carcinoma treated by local excision or subjects with malignancies who have been adequately treated and, in the opinion of the oncologist, have an excellent chance of cancer-free survival Pregnant or nursing women Males with a female partner who is pregnant History of alcohol/drug abuse or dependence within 6 months of the study start (unless participating in a controlled rehabilitation programme) Treatment with an investigational drug or IFN within 30 days or 5 half-lives (whichever is longer) of the screening visit History of platelet clumping that prevents reliable measurement of platelet counts History of major organ transplantation with an existing functional graft Thyroid dysfunction not adequately controlled Subjects planning to have cataract surgery Evidence of portal vein thrombosis on abdominal imaging within 3 months of the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (195):
- United States (52):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Lynwood, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Clemente, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Mateo, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Kinston, North Carolina
  - GSK Investigational Site, Morganton, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Mountain Home, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
- Australia (10):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Brazil (2):
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (9):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Egypt (3):
  - GSK Investigational Site, Al Mansurah
  - GSK Investigational Site, Cairo
  - GSK Investigational Site, Shebeen El-Kom, Menoufeya
- France (11):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (35):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Deggendorf, Bavaria
  - GSK Investigational Site, Hof/Saale, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Beeskow, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Rotenburg (Wümme), Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Leverkusen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Rio, Patras
  - GSK Investigational Site, Thessaloniki
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
- Israel (7):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Nazareth
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (10):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, San Giovanni Rotondo (FG), Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Palermo, Sicily
- GSK Investigational Site, Lahore, Pakistan
- Poland (6):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Racibórz
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, St.Peterburg
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (11):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Taiwan (6):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Chia-Yi Hsien
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taiyuan Hsien
- Ukraine (3):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Saleh MI, Obeidat AR, Anter HA, Khanfar AA. Eltrombopag dose predictors in thrombocytopenic subjects with hepatitis C virus infection. Clin Exp Pharmacol Physiol. 2015 Oct;42(10):1030-5. doi: 10.1111/1440-1681.12451. PMID 26173631
- [Derived] Giannini EG, Afdhal NH, Sigal SH, Muir AJ, Reddy KR, Vijayaraghavan S, Elkashab M, Romero-Gomez M, Dusheiko GM, Iyengar M, Vasey SY, Campbell FM, Theodore D. Non-cirrhotic thrombocytopenic patients with hepatitis C virus: Characteristics and outcome of antiviral therapy. J Gastroenterol Hepatol. 2015 Aug;30(8):1301-8. doi: 10.1111/jgh.12942. PMID 25777337
- [Derived] Afdhal NH, Dusheiko GM, Giannini EG, Chen PJ, Han KH, Mohsin A, Rodriguez-Torres M, Rugina S, Bakulin I, Lawitz E, Shiffman ML, Tayyab GU, Poordad F, Kamel YM, Brainsky A, Geib J, Vasey SY, Patwardhan R, Campbell FM, Theodore D. Eltrombopag increases platelet numbers in thrombocytopenic patients with HCV infection and cirrhosis, allowing for effective antiviral therapy. Gastroenterology. 2014 Feb;146(2):442-52.e1. doi: 10.1053/j.gastro.2013.10.012. Epub 2013 Oct 12. PMID 24126097

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of enrolled participants in the protocol record (n=759) reflects the number of participants randomized to double-blind treatment after completing the Open-label Phase.
Groups:
- Eltrombopag: Open-label Phase: Participants with a platelet count of <75 giga (10^9) cells per liter (Gi/L) initially received eltrombopag 25 milligrams (mg) once daily (QD) for 2 weeks. After 2 weeks, if the platelet count was <100 Gi/L, participants underwent dose escalation to 50 mg QD for 2 weeks. If platelet counts still remained <100 Gi/L, further dose escalations to 75 mg QD (up to 2 weeks) and 100 mg QD (up to a maximum of 3 weeks) were allowed. Participants who achieved platelet counts >=100 Gi/L during the Open-label Phase (maximum of up to 9 weeks) were eligible to enter the Double-blind (DB) Antiviral Treatment Phase, whereas those who failed to reach platelet counts >=100 Gi/L were discontinued from eltrombopag and had to attend the post-treatment follow-up visits.
- Placebo+Antiviral Therapy: DB Phase: Participants completing the OL Phase were administered matching placebo tablets QD in combination with antiviral therapy (peginterferon alfa-2b and ribavirin) for a duration of either 24 or 48 weeks (for participants with Genotype 2/3) or 48 weeks (for participants with Non-Genotype 2/3).
- Eltrombopag+Antiviral Therapy: DB Phase: Participants completing the OL Phase continued on the same dose of eltrombopag received in the OL Phase (dose that effectively raised platelets to >=100 Gi/L) in combination with antiviral therapy (peginterferon alfa-2b and ribavirin) for a duration of either 24 or 48 weeks (for participants with Genotype 2/3) or 48 weeks (for participants with Non-Genotype 2/3).
Period: Open-label Pre-Antiviral Treatment Phase
Arm/Group | Eltrombopag: Open-label Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Started | 805 | 0 | 0
Completed | 759 | 0 | 0
Not Completed | 46 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lost to Follow-up | 12 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0
Not completed — Insufficient Platelet Response | 13 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: Double-bilnd Antiviral Treatment Phase
Arm/Group | Eltrombopag: Open-label Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Started | 0 | 253 | 506
Completed | 0 | 205 | 404
Not Completed | 0 | 48 | 102
Not completed — Adverse Event | 0 | 10 | 27
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 15 | 48
Not completed — Physician Decision | 0 | 5 | 8
Not completed — Withdrawal by Subject | 0 | 17 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase | Total
Number analyzed (Participants) | 253 | 506 | 759
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all randomized participants in the Double-blind (DB) Phase of the study.
  Years | 52.0 (9.15) | 52.4 (8.61) | 52.3 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all randomized participants in the Double-blind (DB) Phase of the study.
  Participants
    Female | 93 | 185 | 278
    Male | 160 | 321 | 481
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study.
  participants
    African American (A)/African | 4 | 8 | 12
    American Indian or Alaska Native | 0 | 1 | 1
    White (W) | 188 | 388 | 576
    Central/South Asian | 16 | 43 | 59
    Japanese/East Asian /South East Asian | 45 | 64 | 109
    American Indian or Alaska Native and White | 0 | 1 | 1
    African A/African and A Indian/Alaska Native and W | 0 | 1 | 1
Number of participants categorized into the indicated genotype for Hepatitic C Virus (HCV) [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. The HCV is a small, enveloped, single-stranded, positive-sense ribonucleic acid (RNA) virus. There are seven major genotypes of HCV, which are indicated numerically from Genotype 1 to 7.
  participants
    Genotype 1 | 160 | 320 | 480
    Genotype 2 | 28 | 40 | 68
    Genotype 3 | 47 | 113 | 160
    Genotype 4 | 17 | 30 | 47
    Genotype 5 | 0 | 0 | 0
    Genotype 6 | 0 | 1 | 1
    Genotype 7 | 0 | 0 | 0
    Missing | 1 | 2 | 3
Number of participants categorized into the indicated Child-Pugh (CP) Class [Number; unit: participants] — The CP score (ranging from 5 to 15, with 5 being mild and 15 being severe), calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess the severity of liver disease. A CP score of 5-6 = Class A (mild), 7-9 = Class B (moderate), and >=10 = Class C (severe).
  participants
    Class A | 242 | 487 | 729
    Class B | 11 | 17 | 28
    Class C | 0 | 0 | 0
    Missing | 0 | 2 | 2
Number of participants with or without previous interferon (IFN) use [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. Participants at Baseline were classified as not having used IFN previously (Naïve) or having used IFN previously (Experienced).
  participants
    Naïve | 182 | 347 | 529
    Experienced | 71 | 159 | 230
Number of participants with the indicated FibroTest/Acti Test (FibroSURE) score [Number; unit: participants] — FibroSURE is a noninvasive blood test that combines the quantitative results of 6 serum biochemical markers (α2-macroglobulin, haptoglobin, apolipoprotein A1, bilirubin, γ-glutamyl transpeptidase [GGT], and ALT) with a participant's age and gender to generate a measure of liver fibrosis/cirrhosis and necroinflammatory activity. It provides a numerical quantitative estimate of liver fibrosis ranging from 0.00 to 1.00, corresponding to the Metavir scoring system of stages F0 to F4 (F0, no fibrosis [F]; F1, portal F; F2, bridging F with few septa; F3, bridging F with many septa; F4=cirrhosis).
  participants
    Score: F0/F1/F2 | 19 | 46 | 65
    Score: F3/F4 | 199 | 405 | 604
    Missing | 35 | 55 | 90
Number of participants with normal or elevated Baseline values for Alanine Aminotransferase (ALT) [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. The normal range of ALT is 0 to 48 International Units per Liter (IU/L).
  participants
    Normal | 49 | 113 | 162
    Elevated | 204 | 393 | 597
Baseline HCV Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: International Units per milliliter] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. HCV RNA was assessed at baseline of the DB Phase. Data are missing for three participants in the Eltrombopag+Antiviral Therapy treatment group.
  International Units per milliliter | 1656788.0 (2564763.45) | 1702729.6 (3066411.11) | 1687415.8 (2907191.97)
Baseline Platelet Count [Mean (Standard Deviation); unit: Giga (10^9) cells per liter (Gi/L)] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. Platelet count eligibility was confirmed at the Baseline visit, prior to administration of eltrombopag, and was defined as the average of the screening and baseline counts, which must be <75 Gi/L.
  Giga (10^9) cells per liter (Gi/L) | 56.56 (13.571) | 56.85 (13.311) | 56.75 (13.390)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR) in the Double-blind (DB) Antiviral Treatment Phase
Description: Participants with SVR are defined as those with non-detectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) at the end of treatment and all subsequent planned visits up to 24 weeks post-completion of the treatment period of the DB Phase.
Time Frame: From Baseline up to Week 48 or Week 72 (for participants with Genotype 2/3) or up to Week 72 (for participants with Non-Genotype 2/3)
Population: Intent-to-Treat (ITT) Population: all participants randomized in the DB Phase
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants | 32 | 97
Statistical Analysis 1: Comparison: Placebo+Antiviral Therapy: DB Phase vs Eltrombopag+Antiviral Therapy: DB Phase; Test type: Superiority or Other; p = 0.0202, Cochran-Mantel-Haenszel — Stratified Cochran-Mantel-Haenszel (CMH) chi-square test adjusted for the randomization strata; Percentage difference in SVR = 6.0, 95% CI 2-sided [1.2 to 10.9] — The estimated value reflects the percentage of participants with SVR in the eltrombopag group minus the percentage of participants with SVR in the placebo group. Adjusted for the actual strata: HCV genotype, baseline platelet count, and HCV RNA

2. Secondary Outcome: Number of Participants Whose Platelet Count Increased From a Baseline Count of <75 Gi/L to a Count Greater Than or Equal to (>=) 100 Giga (10^9) Cells Per Liter (Gi/L) During the Open-label (OL) Pre-Antiviral Treatment Phase
Description: Participants were assessed for a shift from a baseline platelet count of <75 Gi/L to a count >=100 Gi/L during the OL Phase (up to 9 weeks). Local laboratories were used for platelet function tests. Platelet counts were measured by blood draw.
Time Frame: From Baseline up to Week 9 in the OL Phase
Population: Safety Population: all participants who had received study drug in the OL Phase
Measure: Number; unit: participants
Groups:
- Eltrombopag: OL Phase: Participants with a platelet count of <75 giga (10^9) cells per liter (Gi/L) initially received eltrombopag 25 milligrams (mg) once daily (QD) for 2 weeks. After 2 weeks, if the platelet count was <100 Gi/L, participants underwent dose escalation to 50 mg QD for 2 weeks. If platelet counts still remained <100 Gi/L, further dose escalations to 75 mg QD (up to 2 weeks) and 100 mg QD (up to a maximum of 3 weeks) were allowed. Participants who achieved platelet counts >=100 Gi/L during the OL Phase (maximum of up to 9 weeks) were eligible to enter the Double-blind (DB) Antiviral Treatment Phase, whereas those who failed to reach platelet counts >=100 Gi/L were discontinued from eltrombopag and had to attend the post-treatment follow-up visits.
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 805
participants | 773

3. Secondary Outcome: Number of Participants Receiving the Indicated Doses of Eltrombopag in the OL Phase Who Initiated Antiviral Therapy (Peginterferon Alfa-2a and Ribavirin) in the DB Phase
Description: In the OL Phase, participants initially received the lowest dose of eltrombopag (25 mg QD) for 2 weeks. If after this time the platelet count was <100 Gi/L, participants underwent sequential dose escalation to the next highest dose (50 mg QD for up to 2 weeks), with further dose escalations to 75 mg QD (up to 2 weeks) and 100 mg QD (up to a maximum of 3 weeks) if platelet counts remained <100 Gi/L. Participants who achieved platelet counts >=100 Gi/L when receiving any of the eltrombopag doses in the OL Phase initiated antiviral therapy in the DB Phase.
Time Frame: From Baseline up to Week 9 in the OL Phase
Population: Safety Population. Participants with a platelet count >=100 Gi/L and who initiated antiviral therapy during the DB Phase were analyzed.
Measure: Number; unit: participants
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 759
participants
  25 mg | 443
  50 mg | 208
  75 mg | 77
  100 mg | 31

4. Secondary Outcome: Median Platelet Count at the Indicated Time Points During the OL Phase
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts. The Last On Treatment assessment refers to the actual last treatment assessment, not necessarily to the End of Treatment assessment entered by the Investigator.
Time Frame: OL Phase: Baseline; Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, and 9; Antiviral Baseline (up to Week 10); End of Treatment (up to Week 48); 4-week Follow-up (FU) (up to Week 62); 12-week FU (up to Week 70); and 24-week FU (up to Week 82)
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 797
Gi/L
  Baseline, n=797 | 59.0 [12 to 95]
  Day 1, n=714 | 58.0 [5 to 117]
  Week 1, n=791 | 77.0 [5 to 223]
  Week 2, n=530 | 93.0 [9 to 489]
  Week 3, n=288 | 89.0 [10 to 504]
  Week 4, n=161 | 90.0 [10 to 280]
  Week 5, n=98 | 92.0 [9 to 252]
  Week 6, n=55 | 86.0 [14 to 138]
  Week 7, n=35 | 78.0 [11 to 136]
  Week 8, n=24 | 87.5 [15 to 146]
  Week 9, n=4 | 85.5 [66 to 107]
  Antiviral Baseline, n=48 | 131.5 [76 to 274]
  End of Treatment/Withdrawal, n=22 | 76.5 [13 to 257]
  Last on Treatment, n=39 | 87.0 [13 to 267]
  Week 4 Follow-Up, n=20 | 42.0 [11 to 156]
  Week 12 Follow-Up, n=15 | 43.0 [8 to 91]
  Week 24 Follow-Up, n=14 | 41.0 [13 to 87]

5. Secondary Outcome: Median Platelet Count at the Indicated Time Points During the DB Phase
Description: as for outcome 4
Time Frame: DB Phase: Baseline; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44; End of Treatment (up to Week 48); 4-week Follow-up (FU) (up to Week 52); 12-week FU (up to Week 60); and 24-week FU (up to Week 72)
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 252 | 505
Gi/L
  Baseline, n=238, 460 | 140.0 [63 to 365] | 136.0 [43 to 400]
  Week 1, n=247, 494 | 120.0 [42 to 366] | 116.0 [46 to 466]
  Week 2, n=244, 492 | 89.5 [27 to 318] | 124.0 [38 to 553]
  Week 4, n=228, 487 | 51.0 [20 to 180] | 105 [19 to 389]
  Week 6, n=206, 473 | 49.5 [20 to 200] | 100.0 [22 to 417]
  Week 8, n=192, 473 | 50.0 [10 to 191] | 100.0 [19 to 486]
  Week 12, n=176, 451 | 49.7 [21 to 264] | 104.0 [10 to 444]
  Week 16, n=145, 405 | 48.0 [20 to 262] | 102.0 [13 to 365]
  Week 20, n=134, 378 | 50.0 [23 to 257] | 103.0 [21 to 373]
  Week 24, n=99, 263 | 49.0 [19 to 200] | 102.0 [18 to 448]
  Week 28, n=74, 212 | 52.5 [22 to 193] | 102.0 [20 to 355]
  Week 32, n=67, 199 | 49.0 [22 to 195] | 107.0 [14 to 295]
  Week 36, n=63, 185 | 50.0 [16 to 198] | 106.0 [29 to 268]
  Week 40, n=58, 174 | 53.7 [19 to 195] | 106.5 [10 to 351]
  Week 44, n=59, 168 | 53.0 [26 to 197] | 108.7 [26 to 330]
  End of Treatment/Withdrawal, n=240, 468 | 51.0 [10 to 275] | 106.5 [10 to 445]
  Last on Treatment, n=253, 505 | 50.0 [17 to 300] | 105.0 [10 to 330]
  4 week follow up, n=221, 424 | 63.0 [4 to 225] | 89.0 [12 to 333]
  12 week follow up, n=209, 430 | 57.0 [15 to 285] | 62.0 [8 to 280]
  24 week follow up, n=201, 395 | 57.0 [8 to 231] | 59.0 [4 to 297]

6. Secondary Outcome: Number of Participants in the Indicated Categories for Minimum Platelet Count With Antiviral Therapy
Description: The minimum platelet count with antiviral therapy was categorized as follows: <25 Gi/L; >=25 to <50 Gi/L; >=50 to <90 Gi/L; >=90 to <150 Gi/L; >=150 Gi/L to <200 Gi/L; >=200 Gi/L to <400 Gi/L; and >=400 Gi/L.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  <25 Gi/L | 34 | 20
  >=25 to <50 Gi/L | 159 | 76
  >=50 to <90 Gi/L | 49 | 263
  >=90 to <150 Gi/L | 10 | 135
  >=150 to <200 Gi/L | 0 | 8
  >=200 to <400 Gi/L | 0 | 4
  >=400 Gi/L | 0 | 0
  Missing | 1 | 0

7. Secondary Outcome: Number of Participants With Rapid Virological Response (RVR) and Extended RVR (eRVR) During the DB Phase
Description: RVR is defined as the absence of detectable HCV RNA after 4 weeks of antiviral treatment. eRVR is defined as the absence of detectable HCV RNA after 4 weeks of antiviral treatment that persisted through Week 12.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  RVR | 34 | 78
  eRVR | 27 | 69

8. Secondary Outcome: Number of Participants With Early Virological Response (EVR) and Complete EVR (cEVR) During the DB Phase
Description: EVR is defined as a clinically significant reduction from Baseline in HCV RNA (>=2 log10 drop or undetectable) after 12 weeks of antiviral treatment. cEVR is defined as undetectable HCV RNA after 12 weeks of antiviral treatment.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  EVR | 103 | 313
  cEVR | 57 | 174

9. Secondary Outcome: Number of Participants With End of Treatment Response (ETR) and Sustained Virological Response at Week 12 of Follow-up (SVR12) During the DB Phase
Description: ETR is defined as the absence of detectable HCV RNA at the end of antiviral treatment. SVR12 is defined as the absence of detectable HCV RNA at the end of antiviral treatment and the 12-week follow-up assessment.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  ETR | 59 | 190
  SVR12 | 29 | 106

10. Secondary Outcome: Number of Participants in the Indicated Categories for Antiviral Therapy Dose Reductions in the DB Phase
Description: Participants were assigned a score equal to the number of times their dose of antiviral therapy (peginterferon or ribavirin) was reduced (0=no dose reductions [DRs]; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). When possible, every effort was made to maintain the recommended dose of antiviral therapy for the treatment duration in the DB Phase. However, when dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of peginterferon and ribavirin.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  0 | 68 | 231
  1 | 76 | 101
  2 | 40 | 75
  3 | 34 | 47
  >3 | 35 | 52

11. Secondary Outcome: Time to First Dose Reduction of Peginterferon Alfa-2a and Ribavirin Therapy in the DB Phase
Description: Time to first dose reduction was calculated as the time period from the first dose to the first dose reduction.
Time Frame: as for outcome 1
Population: ITT Population. Only those participants with dose reductions were analyzed.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 171 | 208
weeks
  Peginterferon alfa-2a dose reduction, n=171, 208 | 6.58 (7.336) | 10.64 (9.305)
  Ribavirin dose reduction, n=79, 189 | 12.43 (9.681) | 10.99 (8.984)

12. Secondary Outcome: Number of Participants With the Indicated Levels of Peginterferon Dose Reductions in the DB Phase
Description: The assigned dose in the DB Phase of peginterferon alfa-2a was 180 micrograms (µg). For peginterferon dose modification, downward adjustments in one-level increments were considered. The lowest dose of peginterferon alfa-2a that was allowed to be administered was 45 µg. When dose adjustment was required for moderate to severe adverse reactions (clinical and/or laboratory), an initial dose reduction to 135 µg was generally adequate. In some cases, a dose reduction to 90 µg or 45 µg was necessary. Dose increases toward the original dose were considered when the adverse reaction was resolved.
Time Frame: as for outcome 1
Population: ITT Population. One participant could have had more than one dose reduction.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants
  <=25% | 44 | 89
  >25% to <=34% | 33 | 35
  >34% to <=50% | 115 | 112
  >50% | 33 | 30

13. Secondary Outcome: Number of Participants Who Prematurely Discontinued Antiviral Therapy in the DB Phase
Description: The following participants were considered to have discontinued antiviral therapy: participants who were lost to follow-up; participants who withdrew for any reason; participants who died; participants who otherwise did not complete their planned course of antiviral therapy for any reason. The planned duration of antiviral therapy was 48 weeks for participants with Non-Genotype 2/3 and 24 or 48 weeks for participants with Genotype 2/3.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 253 | 506
participants | 164 | 242

14. Secondary Outcome: Number of Participants Categorized as Responders (R) and Non-responders (NR) for SVR and RVR to Antiviral Therapy in the Indicated Variants of Interleukin 28B (IL28B) (or Interferon, Lambda 3)
Description: There are two genetic variants (rs12979860 and rs8099917) mapping near IL28B associated with both interferon-induced SVR and spontaneous HCV clearance. IL28B genotype distribution by response to antiviral therapy (SVR/RVR responders: those who achieved SVR/RVR; SVR/RVR non-responders: those who did not achieve SVR/RVR) was assessed. The effect of genotype was tested by comparing participants that carried 2 copies of the IL28B favorable response allele versus the others (recessive model). Genotypes at rs12979860 were coded as: CC=1, CT or TT=0; rs8099917 was coded as TT=1, GT or GG=0.
Time Frame: as for outcome 1
Population: Pharmacogenetic (PGx) Sub-Population: participants enrolled in this study who provided written informed consent for PGx research with a blood sample for genotyping and who were successfully genotyped for at least one of the two genetic markers under study. Only those participants who were analyzed for SVR and RVR were considered.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 105 | 205
participants
  SVR, rs12979860 (CC), R; n=12, 50 | 10 | 28
  SVR, rs12979860 (CC), NR; n=105, 205 | 24 | 58
  SVR, rs12979860 (CT), R; n=12, 50 | 2 | 18
  SVR, rs12979860 (CT), NR; n=105, 205 | 60 | 111
  SVR, rs12979860 (TT), R; n=12, 50 | 0 | 4
  SVR, rs12979860 (TT), NR; n=105, 205 | 21 | 36
  SVR, rs8099917 (TT), R; n=12, 50 | 11 | 36
  SVR, rs8099917 (TT), NR; n=105, 205 | 48 | 89
  SVR, rs8099917 (GT), R; n=12, 50 | 1 | 13
  SVR, rs8099917 (GT), NR; n=105, 205 | 51 | 99
  SVR, rs8099917 (GG), R; n=12, 50 | 0 | 1
  SVR, rs8099917 (GG), NR; n=105, 205 | 6 | 17
  RVR, rs12979860 (CC), R; n=11, 33 | 6 | 21
  RVR, rs12979860 (CC), NR; n=106, 222 | 28 | 65
  RVR, rs12979860 (CT), R; n=11, 33 | 5 | 11
  RVR, rs12979860 (CT), NR; n=106, 222 | 57 | 118
  RVR, rs12979860 (TT), R; n=11, 33 | 0 | 1
  RVR, rs12979860 (TT), NR; n=106, 222 | 21 | 39
  RVR, rs8099917 (TT), R, n=11, 33 | 9 | 28
  RVR, rs8099917 (TT), NR; n=106, 222 | 50 | 97
  RVR, rs8099917 (GT), R; n=11, 33 | 2 | 5
  RVR, rs8099917 (GT), NR; n=106, 222 | 50 | 107
  RVR, rs8099917 (GG), R; n=11, 33 | 0 | 0
  RVR, rs8099917 (GG), R; n=106, 222 | 6 | 18

15. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline (BL) in Severity Grades for Clinical Chemistry Parameters (Calcium, Glucose [Glu.], Potassium [Pot.], and Sodium [Sod.]), Per Division of Acquired Immunodeficiency Syndrome (DAIDS)
Description: Blood samples for the assessment of clinical chemistry parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL during the DB Phase are reported, per severity grades by DAIDS, for levels of calcium (low=hypocalcemia; high=hypercalcemia), glu. (low=hypoglycemia; high=hyperglycemia), pot. (low=hypokalemia; high=hyperkalemia), and sod. (low=hyponatremia; high=hypernatremia). Per the DAIDS toxicity table, the grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: as for outcome 1
Population: Safety DB Population: all randomized participants who had received study drug in the DB Phase
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 252 | 506
participants
  Calcium (hypocalcemia), Any Grade Increase | 184 | 374
  Calcium (hypocalcemia), Increase to G1 | 140 | 246
  Calcium (hypocalcemia), Increase to G2 | 42 | 122
  Calcium (hypocalcemia), Increase to G3 | 2 | 4
  Calcium (hypocalcemia), Increase to G4 | 0 | 2
  Calcium (hypercalcemia), Any Grade Increase | 2 | 1
  Calcium (hypercalcemia), Increase to G1 | 1 | 1
  Calcium (hypercalcemia), Increase to G2 | 1 | 0
  Calcium (hypercalcemia), Increase to G3 | 0 | 0
  Calcium (hypercalcemia), Increase to G4 | 0 | 0
  Glu. (hypoglycemia), Any Grade Increase | 31 | 90
  Glu. (hypoglycemia), Increase to G1 | 17 | 45
  Glu. (hypoglycemia), Increase to G2 | 10 | 31
  Glu. (hypoglycemia), Increase to G3 | 4 | 9
  Glu. (hypoglycemia), Increase to G4 | 0 | 5
  Glu. (hyperglycemia), Any Grade Increase | 128 | 277
  Glu. (hyperglycemia), Increase to G1 | 31 | 68
  Glu. (hyperglycemia), Increase to G2 | 77 | 161
  Glu. (hyperglycemia), Increase to G3 | 19 | 44
  Glu. (hyperglycemia), Increase to G4 | 1 | 4
  Pot. (hyperkalemia), Any Grade Increase | 3 | 15
  Pot. (hyperkalemia), Increase to G1 | 2 | 7
  Pot. (hyperkalemia), Increase to G2 | 1 | 3
  Pot. (hyperkalemia), Increase to G3 | 0 | 2
  Pot. (hyperkalemia), Increase to G4 | 0 | 3
  Pot. (hypokalemia), Any Grade Increase | 53 | 74
  Pot. (hypokalemia), Increase to G1 | 48 | 66
  Pot. (hypokalemia), Increase to G2 | 5 | 6
  Pot. (hypokalemia), Increase to G3 | 0 | 2
  Pot. (hypokalemia), Increase to G4 | 0 | 0
  Sod. (hypernatremia), Any Grade Increase | 14 | 21
  Sod. (hypernatremia), Increase to G1 | 14 | 20
  Sod. (hypernatremia), Increase to G2 | 0 | 1
  Sod. (hypernatremia), Increase to G3 | 0 | 0
  Sod. (hypernatremia), Increase to G4 | 0 | 0
  Sod. (hyponatremia), Any Grade Increase | 72 | 128
  Sod. (hyponatremia), Increase to G1 | 69 | 118
  Sod. (hyponatremia), Increase to G2 | 3 | 8
  Sod. (hyponatremia), Increase to G3 | 0 | 1
  Sod. (hyponatremia), Increase to G4 | 0 | 1

16. Secondary Outcome: Number of Participants With the Indicated Shifts From BL in Severity Grades for for Hematology Parameters (Hemoglobin, Lymphocytes [Lym.], Total Neutrophils [Tot Neu.], and White Blood Cells [WBC]), Per DAIDS
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL during the DB Phase are reported, per severity grades by DAIDS, for levels of hemoglobin (low=anemia), lymphocytes (low=lymphocytopenia), total neutrophils (low=neutropenia), and white blood cells (low=leukocytopenia). Per the DAIDS toxicity table, grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: as for outcome 1
Population: Safety DB Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 252 | 506
participants
  Hemoglobin (anemia), Any Grade Increase | 161 | 361
  Hemoglobin (anemia), Increase to G1 | 46 | 112
  Hemoglobin (anemia), Increase to G2 | 64 | 129
  Hemoglobin (anemia), Increase to G3 | 48 | 114
  Hemoglobin (anemia), Increase to G4 | 3 | 6
  Lym. (lymphocytopenia), Any Grade Increase | 136 | 346
  Lym. (lymphocytopenia), Increase to G1 | 16 | 43
  Lym. (lymphocytopenia), Increase to G2 | 38 | 80
  Lym. (lymphocytopenia), Increase to G3 | 48 | 109
  Lym. (lymphocytopenia), Increase to G4 | 34 | 114
  Tot Neu. (neutropenia), Any Grade Increase | 208 | 394
  Tot Neu. (neutropenia), Increase to G1 | 50 | 106
  Tot Neu. (neutropenia), Increase to G2 | 53 | 113
  Tot Neu. (neutropenia), Increase to G3 | 73 | 128
  Tot Neu. (neutropenia), Increase to G4 | 32 | 47
  WBC (leukocytopenia), Any Grade Increase | 191 | 391
  WBC (leukocytopenia), Increase to G1 | 56 | 113
  WBC (leukocytopenia), Increase to G2 | 69 | 145
  WBC (leukocytopenia), Increase to G3 | 58 | 110
  WBC (leukocytopenia), Increase to G4 | 8 | 23

17. Secondary Outcome: Number of Participants in the Indicated Categories for Cataract Event During the DB Phase, Per Clinical Events Committee (CEC) Adjudication
Description: Ophthalmic (pertaining to eye) assessments were performed during the study. A cataract event is defined as an event ascertained to be a cataract (opacity or cloudiness of the lens of the eye, causing impairment of vision) by at least one of the CEC members (comprised of expert ophthalmologists who provided objective medical review of the blinded ophthalmic data). Per the CEC, cataract events were categorized as: (1) Cataract Progression (CP; progression of cataracts present at BL); and (2) Incident Cataract (IC; development of new cataracts). One eye=unilateral; both eyes=bilateral.
Time Frame: as for outcome 1
Population: Safety DB Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 252 | 506
participants
  Unilateral CP, Genotype 2/3 | 0 | 1
  Unilateral CP, Non-genotype 2/3 | 4 | 6
  Bilateral CP, Genotype 2/3 | 3 | 1
  Bilateral CP, Non-genotype 2/3 | 1 | 7
  Unilateral IP, Genotype 2/3 | 1 | 4
  Unilateral IP, Non-genotype 2/3 | 1 | 6
  Bilateral IP, Genotype 2/3 | 3 | 1
  Bilateral IP, Non-genotype 2/3 | 3 | 10

18. Secondary Outcome: Number of Participants Assessed as Normal and Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) at the Indicated Time Points During the DB Phase
Description: Duplicate 12-lead ECGs were required at Screening/BL, Antiviral BL, and at 12 weekly intervals during the study. The number of participants with an ECG status of normal, abnormal, CS, or NCS, as determined by the Investigator, was reported. Normal, all ECG parameters within accepted normal ranges. Abnormal, ECG finding(s) outside of normal ranges. CS, ECG with a CS abnormality that meets exclusion criteria. NCS, ECG with an abnormality not CS or meeting exclusion criteria, per Investigator, based on reasonable standards of clinical judgment.
Time Frame: DB Phase: Antiviral BL (up to Week 10); End of Treatment (up to Week 52); and 24-week FU (up to Week 72)
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 252 | 505
participants
  Antiviral BL, Normal, n=232, 478 | 147 | 332
  Antiviral BL, Abnormal - NCS, n=232, 478 | 63 | 103
  Antiviral BL, Abnormal - CS, n=232, 478 | 22 | 43
  End of Treatment, Normal, n=218, 428 | 134 | 291
  End of Treatment, Abnormal - NCS, n=218, 428 | 62 | 103
  End of Treatment, Abnormal - CS, n=218, 428 | 22 | 34
  24-week FU, Normal, n=194, 383 | 123 | 238
  24-week FU, Abnormal - NCS, n=194, 383 | 49 | 107
  24-week FU, Abnormal - CS, n=194, 383 | 22 | 38
  Worst ECG post-BL, Normal, n=252, 505 | 113 | 233
  Worst ECG post-BL, Abnormal - NCS, n=252, 505 | 91 | 171
  Worst ECG post-BL, Abnormal - CS, n=252, 505 | 48 | 101

19. Secondary Outcome: Number of Participants With CS and NCS Change From Baseline for 12-lead ECG at the Indicated Time Points During the DB Phase
Description: Duplicate 12-lead ECGs were required at Screening/BL, Antiviral BL, and at 12 weekly intervals during the study. The number of participants with a CS and a NCS change from baseline in ECG status, as determined by the Investigator, was reported. CS, ECG with a CS abnormality that meets exclusion criteria. NCS, ECG with an abnormality not CS or meeting exclusion criteria, per Investigator, based on reasonable standards of clinical judgment. "Not applicable" indicates that information was not provided by the investigator on whether the change from baseline ECG was CS or NCS.
Time Frame: End of Treatment (up to Week 52); and 24-week FU (up to Week 72)
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 218 | 428
participants
  End of Treatment, CS change from BL, n=218, 428 | 0 | 7
  End of Treatment, NCS change from BL, n=218, 428 | 218 | 420
  End of Treatment, Not applicable, n=218, 428 | 0 | 1
  24-week FU, CS change from BL, n=194, 383 | 1 | 4
  24-week FU, NCS change from BL, n=194, 383 | 193 | 379

20. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points During the DB Phase
Description: Participant's blood pressure was measured at the indicated time points during the study. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic blood pressure is a measure of blood pressure while the heart is relaxed. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 246 | 494
Millimeters of mercury (mmHg)
  SBP, Week 1, n=246, 491 | -3.00 (13.541) | -2.36 (12.296)
  SBP, Week 2, n=242, 494 | -3.25 (13.800) | -3.74 (13.122)
  SBP, Week 4, n=228, 485 | -3.75 (13.781) | -3.91 (13.780)
  SBP, Week 6, n=206, 471 | -3.36 (14.405) | -3.85 (14.624)
  SBP, Week 8, n=190, 472 | -2.72 (14.073) | -4.33 (14.401)
  SBP, Week 12, n=175, 452 | -2.16 (15.297) | -4.30 (14.377)
  SBP, Week 16, n=143, 403 | -3.16 (15.426) | -4.59 (13.579)
  SBP, Week 20, n=133, 374 | -2.50 (14.387) | -4.12 (14.908)
  SBP, Week 24, n=99, 263 | -1.97 (14.820) | -3.94 (14.917)
  SBP, Week 28, n=74, 211 | -0.69 (14.663) | -4.99 (14.557)
  SBP, Week 32, n=67, 197 | -1.46 (13.904) | -5.61 (13.523)
  SBP, Week 36, n=62, 186 | -1.31 (13.803) | -4.40 (14.842)
  SBP, Week 40, n=59, 173 | 0.10 (13.605) | -4.31 (13.941)
  SBP, Week 44, n=59, 167 | 0.56 (11.689) | -4.54 (13.794)
  SBP, End of Treatment, n=238, 468 | -2.03 (13.259) | -3.98 (15.318)
  SBP, 4-week FU, n=221, 426 | -1.14 (14.095) | -1.65 (15.122)
  SBP, 12-week FU, n=207, 432 | -0.11 (14.113) | -0.86 (14.806)
  SBP, 24-week FU, n=203, 398 | 1.10 (14.545) | 0.25 (14.518)
  DBP, Week 1, n=246, 491 | -1.43 (9.235) | -1.37 (8.224)
  DBP, Week 2, n=242, 493 | -1.55 (9.217) | -1.86 (8.946)
  DBP, Week 4, n=228, 485 | -1.84 (9.726) | -2.72 (9.467)
  DBP, Week 6, n=206, 471 | -2.16 (8.939) | -2.95 (9.859)
  DBP, Week 8, n=190, 472 | -1.24 (9.517) | -2.68 (9.901)
  DBP, Week 12, n=175, 452 | -1.31 (8.781) | -3.23 (10.025)
  DBP, Week 16, n=143, 403 | -1.54 (9.684) | -3.31 (9.899)
  DBP, Week 20, n=133, 374 | -0.93 (10.582) | -3.08 (9.606)
  DBP, Week 24, n=99, 263 | -1.66 (10.207) | -3.54 (9.313)
  DBP, Week 28, n=74, 211 | -1.23 (9.538) | -3.42 (10.502)
  DBP, Week 32, n=67, 197 | -0.54 (10.445) | -3.76 (9.527)
  DBP, Week 36, n=62, 186 | -0.74 (9.559) | -3.59 (9.211)
  DBP, Week 40, n=59, 173 | 0.34 (9.343) | -3.32 (9.517)
  DBP, Week 44, n=59, 167 | 0.92 (9.033) | -3.77 (10.134)
  DBP, End of Treatment, n=238, 468 | -1.55 (9.174) | -3.59 (10.254)
  DBP, 4-week FU, n=221, 426 | -0.83 (9.102) | -2.20 (9.824)
  DBP, 12-week FU, n=207, 432 | -0.78 (10.253) | -1.76 (9.903)
  DBP, 24-week FU, n=203, 398 | 0.03 (9.814) | -1.61 (9.339)

21. Secondary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points During the DB Phase
Description: Heart rate was measured in participants at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 244 | 490
beats per minute
  Week 1, n=244, 490 | 1.16 (8.358) | -0.43 (8.629)
  Week 2, n=242, 490 | 1.89 (8.510) | 0.78 (9.644)
  Week 4, n=227, 483 | 2.47 (9.464) | 1.50 (9.739)
  Week 6, n=205, 470 | 3.23 (9.158) | 1.19 (8.708)
  Week 8, n=190, 472 | 2.91 (9.751) | 1.78 (9.227)
  Week 12, n=174, 450 | 4.28 (10.188) | 2.02 (9.539)
  Week 16, n=143, 403 | 5.87 (9.975) | 2.38 (10.419)
  Week 20, n=132, 371 | 5.73 (9.688) | 2.10 (9.530)
  Week 24, n=99, 262 | 3.77 (9.912) | 2.03 (9.399)
  Week 28, n=74, 211 | 2.72 (10.038) | 1.64 (10.328)
  Week 32, n=67, 196 | 4.28 (8.281) | 1.62 (9.676)
  Week 36, n=62, 186 | 5.42 (10.109) | 2.11 (10.205)
  Week 40, n=59, 171 | 4.83 (8.919) | 0.78 (9.895)
  Week 44, n=59, 165 | 5.53 (11.005) | 1.16 (8.846)
  End of Treatment, n=237, 467 | 4.01 (10.606) | 2.89 (11.134)
  4-week FU, n=220, 422 | 4.27 (10.432) | 2.11 (10.113)
  12-week FU, n=206, 429 | 1.73 (9.707) | 0.74 (9.955)
  24-week FU, n=202, 395 | 0.14 (9.803) | -1.90 (9.176)

22. Secondary Outcome: Mean Change From Baseline in Weight at the Indicated Time Points During the DB Phase
Description: The weight of participants was recorded at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 248 | 495
Kilograms (kg)
  Week 1, n=248, 492 | -0.65 (2.201) | -0.68 (2.062)
  Week 2, n=244, 495 | -0.88 (1.983) | -1.06 (2.809)
  Week 4, n=229, 488 | -1.30 (2.374) | -1.30 (2.488)
  Week 6, n=207, 476 | -1.42 (2.464) | -1.68 (2.652)
  Week 8, n=191, 473 | -1.89 (2.793) | -2.11 (2.810)
  Week 12, n=175, 453 | -2.18 (2.985) | -2.83 (3.440)
  Week 16, n=145, 406 | -2.37 (3.247) | -3.32 (3.798)
  Week 20, n=134, 378 | -3.08 (3.684) | -3.99 (4.040)
  Week 24, n=99, 265 | -4.04 (4.148) | -4.75 (4.175)
  Week 28, n=74, 212 | -4.57 (4.749) | -5.09 (5.016)
  Week 32, n=67, 200 | -4.50 (4.397) | -5.52 (5.369)
  Week 36, n=63, 188 | -4.54 (4.739) | -5.39 (7.476)
  Week 40, n=59, 174 | -4.99 (4.612) | -5.87 (5.571)
  Week 44, n=59, 168 | -4.79 (5.475) | -5.89 (5.661)
  End of Treatment, n=240, 470 | -3.28 (4.361) | -4.69 (5.180)
  4-week FU, n=223, 425 | -2.78 (4.318) | -3.84 (6.381)
  12-week FU, n=210, 434 | -1.98 (4.088) | -2.99 (5.999)
  24-week FU, n=205, 401 | -1.36 (4.568) | -1.51 (7.683)

23. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI) at the Indicated Time Points During the DB Phase
Description: The BMI for participants was calculated at the indicated time points as body weight in kilograms divided by height in meters squared. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms per meters squared (kg/m^2)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 248 | 493
Kilograms per meters squared (kg/m^2)
  Week 1, n=248, 490 | -0.23 (0.771) | -0.23 (0.713)
  Week 2, n=244, 493 | -0.31 (0.691) | -0.36 (0.921)
  Week 4, n=229, 486 | -0.46 (0.823) | -0.45 (0.855)
  Week 6, n=207, 474 | -0.50 (0.871) | -0.58 (0.893)
  Week 8, n=191, 471 | -0.66 (0.967) | -0.73 (0.955)
  Week 12, n=175, 451 | -0.77 (1.055) | -0.97 (1.167)
  Week 16, n=145, 404 | -0.85 (1.158) | -1.15 (1.285)
  Week 20, n=134, 376 | -1.11 (1.324) | -1.39 (1.377)
  Week 24, n=99, 264 | -1.46 (1.509) | -1.66 (1.624)
  Week 28, n=74, 211 | -1.67 (1.731) | -1.79 (1.733)
  Week 32, n=67, 199 | -1.64 (1.586) | -1.94 (1.844)
  Week 36, n=63, 187 | -1.65 (1.703) | -1.89 (2.651)
  Week 40, n=59, 173 | -1.81 (1.671) | -2.09 (1.953)
  Week 44, n=59, 167 | -1.73 (2.007) | -2.09 (1.942)
  End of Treatment, n=240, 468 | -1.16 (1.553) | -1.64 (1.783)
  4-week FU, n=223, 423 | -0.98 (1.519) | -1.35 (2.306)
  12-week FU, n=210, 432 | -0.70 (1.434) | -1.06 (2.055)
  24-week FU, n=205, 399 | -0.47 (1.544) | -0.53 (2.736)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported for the Double-blind (DB) on-treatment + 30 days period (up to Study Week 52).
Description: In the study, AEs were collected during the Open-Label (OL) Pre-Antiviral Treatment Phase and the Double-Blind (DB) Phase, which included antiviral therapy and a 6-month post-therapy follow-up. Data for SAEs and AEs are presented for the Safety Population, comprised of all randomized participants who received the study drug.
Arm/Group | Eltrombopag: OL Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Serious Adverse Events (participants affected / at risk) | 9/805 | 49/252 | 119/506
Other Adverse Events (participants affected / at risk) | 0/805 | 226/252 | 459/506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag: OL Phase (N=805) | Placebo+Antiviral Therapy: DB Phase (N=252) | Eltrombopag+Antiviral Therapy: DB Phase (N=506)
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 7
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Gastric varices hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7 | 22
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 2 | 6
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 5
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 | 4 | 4
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 3
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Varices esophageal (Gastrointestinal disorders) | 0 | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 4
Cellulitis (Infections and infestations) | 0 | 2 | 2
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 2
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Campylobacter intestinal infection (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Actinomycotic pulmonary infection (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Anogenital warts (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0
Salmonella bacteremia (Infections and infestations) | 0 | 1 | 0
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 1
Generalized edema (General disorders) | 0 | 0 | 1
Induration (General disorders) | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Edema peripheral (General disorders) | 0 | 1 | 1
Sudden death (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 5
Anemia hemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 9
Coma hepatic (Nervous system disorders) | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Osmotic demyelination syndrome (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 2
Abnormal behavior (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 9
Visual acuity reduced (Eye disorders) | 0 | 1 | 2
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal hemorrhage (Eye disorders) | 0 | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Amyloidosis (Immune system disorders) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag: OL Phase (N=805) | Placebo+Antiviral Therapy: DB Phase (N=252) | Eltrombopag+Antiviral Therapy: DB Phase (N=506)
Pyrexia (General disorders) | 0 | 60 | 141
Fatigue (General disorders) | 0 | 53 | 124
Influenza like illness (General disorders) | 0 | 36 | 100
Asthenia (General disorders) | 0 | 28 | 86
Chills (General disorders) | 0 | 32 | 72
Irritability (General disorders) | 0 | 11 | 34
Edema peripheral (General disorders) | 0 | 3 | 36
Injection site erythema (General disorders) | 0 | 14 | 22
Anemia (Blood and lymphatic system disorders) | 0 | 90 | 200
Neutropenia (Blood and lymphatic system disorders) | 0 | 83 | 139
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 83 | 61
Leukopenia (Blood and lymphatic system disorders) | 0 | 32 | 57
Nausea (Gastrointestinal disorders) | 0 | 38 | 92
Diarrhea (Gastrointestinal disorders) | 0 | 24 | 92
Vomiting (Gastrointestinal disorders) | 0 | 18 | 41
Abdominal pain (Gastrointestinal disorders) | 0 | 10 | 31
Abdominal pain upper (Gastrointestinal disorders) | 0 | 13 | 28
Ascites (Gastrointestinal disorders) | 0 | 6 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 34 | 71
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 12 | 50
Rash (Skin and subcutaneous tissue disorders) | 0 | 10 | 38
Headache (Nervous system disorders) | 0 | 50 | 95
Dizziness (Nervous system disorders) | 0 | 13 | 40
Weight decreased (Investigations) | 0 | 17 | 49
White blood cell count decreased (Investigations) | 0 | 18 | 42
Hemoglobin decreased (Investigations) | 0 | 16 | 34
Blood bilirubin increased (Investigations) | 0 | 7 | 36
Platelet count decreased (Investigations) | 0 | 14 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 26 | 64
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 22 | 51
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 20 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 14 | 36
Insomnia (Psychiatric disorders) | 0 | 27 | 72
Depression (Psychiatric disorders) | 0 | 19 | 47
Decreased appetite (Metabolism and nutrition disorders) | 0 | 36 | 94
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 11 | 42
Urinary tract infection (Infections and infestations) | 0 | 13 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.